CLINICAL TRIAL: NCT05193708
Title: Comparison of Bracket Bonding Variables Using Bonding Guide 3D Printed With Fusion Deposition Modeling Versus Digital Indirect Bonding. A Randomized Controlled Trial.
Brief Title: Comparison of Bracket Bonding Variables Using 3D Printed Bonding Guide Versus Digital Indirect Bonding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelhady Nasef, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 777
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-08

CONDITIONS: Dental Bonding; Orthodontic Brackets; Indirect Bonding
Keywords: digital indirect; windowed bonding tray

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital Indirect bonding (Active Comparator): An indirect bonding tray will be fabricated from a 3D printed model
  Interventions: Device: Windowed Bonding
- Windowed Bonding technique (Experimental): 3D printed guide with windows for positioning the bracket
  Interventions: Device: Digital Indirect bonding tray

INTERVENTIONS:
Device: Windowed Bonding — A 3D printed tray/guide with open window for the orthodontic brackets
  Arms: Digital Indirect bonding
Device: Digital Indirect bonding tray — Vacuum formed on a 3d printer cast with brackets
  Arms: Windowed Bonding technique

SUMMARY:
The windowed direct-indirect bonding is a new bonding technique that could provide a simple and cheap method for fast and precise brackets bonding. There are still not enough studies to evaluate the effectiveness of this method in terms of accuracy, bonding time, bonding failure and cost.

This study is designed to answer these questions and compare the forementioned bonding technique with digital indirect bonding and finally provide the clinician a recommendation on the best bonding technique. This study introduces as well a new method of fabrication of the windowed template using Fusion Deposition Modeling (FDM) 3D printing technology.

DETAILED DESCRIPTION:
This study will compare two bonding techniques, the windowed bonding technique and digital indirect bonding. They will be compared regarding accuracy, bonding time, bonding failure and cost. Patients will be selected according to the eligibility criteria, random sequence generation and blind allocation will be performed. ( A randomized clinical trial). Patients will be allocated to one of the groups either the windowed bonding or the digital indirect bonding.

Both groups will undergo similar steps initially. First, the patient's teeth will be digitized using an intraoral scanner. Then using 3 shape software, the model will be prepared and brackets will be positioned virtually on the 3D models. Then, in the windowed bonding technique, the windowed tray will be designed and later 3D printed, while in the digital indirect technique the model with the brackets will be 3D printed and a tray will be fabricated on the model manually.

After the fabrication of the tray, the brackets will be transferred to the patient using the tray or directly bonded using the windowed tray guide.

The patient's teeth will be scanned after bonding and this 3D model will be compared with the initial brackets setup that was made previously on the software.

ELIGIBILITY:
Inclusion Criteria:

* - Patients who need Orthodontic treatment with full dentition excluding 3rd molars.
* Fully erupted 5-5 with normal anatomy.
* The patient's age range is from 12 to 60 years of age.
* Both extraction and non-extraction cases are included.

Exclusion Criteria:

* - Patients with caries, fluorosis, enamel hypoplasia, restorations, or fractures.
* Patients with severe rotations.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2022-10-22 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Bonding accuracy | After bonding immediately
  Deterring the accuracy of bracket position

SECONDARY OUTCOMES:
Bonding time | Time begins starting from etching procedure till the final bracket cured, this will be measured in minutes (~ 20 minutes)
  Calculating the time of bonding

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt